CLINICAL TRIAL: NCT05556005
Title: Effect Of Trimetazidine On Left Ventricular Functions and Inflammatory Markers of Patients With Type 2 Diabetes Mellitus
Brief Title: Efficacy of Trimetazidine in Diabetic Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Heba ibrahim Mohamed serag, Assistant lecturer of clinical pharmacy- faculty of pharmacy, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RHDIRB2020110301
Record Dates: First submitted 2022-09-21; First posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Diabetes Mellitus, Type 2; Diabetic Cardiomyopathies
Keywords: Trimetazidine; Diastolic dysfunction; diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Cardiomyopathies; Diabetes Mellitus | interventions — Trimetazidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): Patients will receive 35 mg of Trimetazidine modified release tablet twice daily in addition to their standard treatment for three months.
  Interventions: Drug: Trimetazidine Dihydrochloride
- Group 2 (Placebo Comparator): Patients will receive Placebo tablet twice daily in addition to their standard treatment for three months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Trimetazidine Dihydrochloride — Trimetazidine Dihydrochloride 35 mg modified release tablet used twice daily
  Other Names: Vasteral mr
  Arms: Group 1
Drug: Placebo — Starch tablets used twice daily
  Arms: Group 2

SUMMARY:
Subclinical diastolic dysfunction represents the early phase of diabetic cardiomyopathy and is a common complication among type 2 diabetic patients that increases mortality rate among those patients and can progress to heart failure with preserved ejection fraction. Trimetazidine is an anti-ischemic agent widely used in the treatment of coronary artery disease and it has positive effects on energy metabolism in heart failure.

Therefore, we hypothesized that trimetazidine may have potential benefit on the amelioration of the inflammatory insult and improving the clinical outcomes in patients with diabetic cardiomyopathy especially if applied in the early stages.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 40-75 years
2. Patients with echocardiographic evidence of grade I or II diastolic dysfunction with LVEF ≥50%

Exclusion Criteria:

1. Patients with valvular, congenital or ischemic heart disease.
2. Patients with inadequately controlled hypertension (blood pressure>140/90 mm Hg)
3. Patients with HbA1c% <10 %
4. Patients with history of intolerance or allergic response to TMZ
5. Patients with severe liver dysfunction or severe renal dysfunction (creatinine clearance < 30 ml/min)
6. Patients with other significant comorbidities such as malignancy, significant psychiatric illness, autoimmune diseases.
7. Patients with Parkinson's disease or motor disorders
8. Pregnancy and breast feeding

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-18 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Left ventricular functions at 3 months | at baseline and after three months of intervention
  assessed using echocardiographic and tissue doppler evaluation

SECONDARY OUTCOMES:
Change from baseline Tumor necrosis factor alpha at 3 months | at baseline and after three months of intervention
  assessed using ELISA technique
Change from baseline Transforming growth factor beta 1 at 3 months | at baseline and after three months of intervention
  assessed using ELISA technique

CONTACTS AND LOCATIONS:
Locations (1):
- Ainshams university hospitals, Cairo, Egypt

REFERENCES:
- [Derived] Serag H, Wakeel LE, William V, Abdelsalam M, Abdelsalam A, Sayed R. Effect of trimetazidine on left ventricular functions and cardiac biomarkers in diabetic patients with left ventricular diastolic dysfunction: a randomized controlled trial. Sci Rep. 2025 Jan 16;15(1):2115. doi: 10.1038/s41598-024-83213-w. PMID 39814796